CLINICAL TRIAL: NCT01458847
Title: A Single Dose, Dose-escalating, Phase I Study to Evaluate Safety, Tolerability and Pharmacokinetics of Intravesical Cis-urocanic Acid (Cis-UCA) in Patients With Primary or Recurrent Non-muscle Invasive Bladder Cancer
Brief Title: Cis-urocanic Acid (Cis-UCA) in Patients With Primary or Recurrent Non-muscle Invasive Bladder Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioCis Pharma Ltd (Industry)
Collaborators: Turku University Hospital (Other Government); Tampere University Hospital (Other); FinnMedi Oy (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL08003; 2009-011287-11 (EudraCT Number)
Record Dates: First submitted 2011-10-04; First posted 2011-10-25 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Non-muscle Invasive Bladder Cancer
Keywords: bladder cancer; cis-urocanic acid; primary; recurrent; non-muscle
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort I: 2% cis-UCA solution (50 ml) (Experimental)
  Interventions: Drug: cis-UCA solution
- Cohort II: 4% cis-UCA solution (50 ml) (Experimental)
  Interventions: Drug: cis-UCA solution
- Cohort III: 6% cis-UCA solution (50 ml) (Experimental)
  Interventions: Drug: cis-UCA solution

INTERVENTIONS:
Drug: cis-UCA solution — Cohort I: 2% cis-UCA solution (50 ml); min 3, max 12 patients
  Arms: Cohort I: 2% cis-UCA solution (50 ml)
Drug: cis-UCA solution — Cohort II: 4% cis-UCA solution (50 ml); min 0, max 12 patients
  Arms: Cohort II: 4% cis-UCA solution (50 ml)
Drug: cis-UCA solution — Cohort III: 6% cis-UCA solution (50 ml); min 0, max 12 patients
  Arms: Cohort III: 6% cis-UCA solution (50 ml)

SUMMARY:
The purpose of this study is to evaluate safety, tolerability and pharmacokinetics of intravesical cis-urocanic acid in patients with primary or recurrent non-muscle invasive bladder cancer.

DETAILED DESCRIPTION:
This is a single dose, dose-escalating, Phase I study to evaluate safety, tolerability and pharmacokinetics of intravesical cis-urocanic acid (cis-UCA) in patients with primary or recurrent non-muscle invasive bladder cancer.

The primary objectives is to evaluate safety and tolerability of cis-UCA after a single intravesical instillation with escalating doses and to determine the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of cis-UCA after a single intravesical instillation with escalating doses.

The secondary objectives are to evaluate pharmacokinetics of cis-UCA after a single intravesical instillation with escalating doses, to obtain preliminary information on possible anti-tumor effects of cis-UCA by cystoscopy and histological evaluation after a single intravesical instillation with escalating doses, and to evaluate the effects of cis-UCA on different surrogate biochemical markers on tumor growth and differentiation after a single intravesical instillation with escalating doses.

The key eligibility criteria are the following: Patients with primary or recurrent non-muscle invasive bladder cancer; eligible for intravesical treatment; age 18-80 years; WHO performance status 0-2; acceptable liver, renal and hematological function within 30 days prior to inclusion.

At minimum 3 patients and at maximum 24 patients is planned to be included in the study. The fixed dose-escalation levels will be used.

Up to three dose cohorts are planned to be included:

* Cohort I: 2% cis-UCA solution (50 ml); min 3, max 12 patients
* Cohort II: 4% cis-UCA solution (50 ml); min 0, max 12 patients
* Cohort III: 6% cis-UCA solution (50 ml); min 0, max 12 patients

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained prior to any screening procedures
2. Patients with primary or recurrent non-muscle invasive bladder cancer
3. The patient is eligible for intravesical instillation
4. Age 18-80 years
5. WHO performance status 0-2
6. Body weight at least 50 kg for males and 45 kg for females; body mass index (BMI) 18-35 kg/m2
7. Diagnostic cystoscopy performed within 30 days prior to screening visit
8. Negative pregnancy test (premenopausal female patients) at screening and use of adequate contraceptive measures (both male and female patients) throughout the study and 30 days after the cis-UCA dose oPremenopausal female volunteers should be either surgically sterile or using a reliable contraception method: intrauterine device (hormonal or non-hormonal); oral combination pill or hormonal contraception patch; or two of the following: intra-vaginal hormonal ring, oral contraceptive containing progestin only, spermicidal foam, condom, sterilization of male sexual partner (surgical vasectomy) oPatients with no current heterosexual relationship may be included according to the judgment of the Investigator oIf menopause occurred 2 years ago at the minimum, no contraception is required for female participants, nor pregnancy tests oReliable contraception for male patients is concordant with above listed methods for females, as applicable
9. Acceptable liver function, renal function and hematological status at screening
10. Urinalysis showing no clinically significant abnormalities except those attributable for bladder cancer

Exclusion Criteria:

1. Previously diagnosed bladder fibrosis
2. Total bladder capacity estimated by cystoscopy to be less that 150 ml
3. Urinary incontinence of that severity that according to the opinion of the Urologist/Investigator would compromise the ability of the patient to retain the study drug intravesical instillation for one hour
4. Severe irritative voiding symptoms, such as urgency, frequency and nocturia that could compromise protocol objectives in the opinion of the Urologist/Investigator
5. Serious disease (e.g., hydronephrosis, renal or liver failure or other condition) that could compromise protocol objectives in the opinion of the Urologist/Investigator
6. Active, uncontrolled bacterial, viral, or fungal infections, including urinary tract infection
7. Previous treatment with radiotherapy, or systemic chemotherapy.
8. Intravesical instillation(s) within 6 months with BCG or cytostatic agents
9. Known allergy to cis-UCA-instillation solution (see Section 5.1 for excipients).
10. Having participated in a clinical study with cis-UCA previously
11. Known any serious immunodeficiency condition
12. Donation of blood or participation in another drug study within 60 days (males) or 90 days (females) before the intravesical instillation in this study
13. Any clinically significant laboratory test result (including positive tests for HIV and hepatitis B or C) according to Investigator/Urologist
14. Excessive use of alcohol (on average more than 24 units per week for males, and more that 16 units per weeks for females; unit = 4 cl spirits or equivalent)
15. Clinically significant illness (except bladder cancer) within 30 days before the screening visit or any other condition, such as vesicourethral reflux (VUR), or complicated urinary stone disease that in the opinion of the Investigator would interfere with the evaluation of the study results or constitute a health hazard for the patient
16. Regular use of urine alkalinizing agents/drugs (e.g., acetazolamide, calcium phosphates, aluminium hydroxide, sodium bicarbonate, sodium carbonate, sodium citrate, potassium citrate) that might interfere with the evaluation of the study results
17. Unwillingness or doubtful capacity to comply with the protocol
18. Doubtful availability, in the opinion of the Investigator, to complete the study
19. Poor peripheral venous access -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Bladder-related AEs | until resection, max 2 months
Urinalysis | participants will be followed until resection, an expected average of 2 months
Evaluation of the appearance of normal bladder epithelium after the cis-UCA dose by cystoscopy during the planned surgical procedure | participants will be followed until resection, an expected average of 2 months
  cystoscopy descriptions

SECONDARY OUTCOMES:
Area Under Curve (AUC) | Predose, 30 min, 45 min, 1 h, 1.5 h, 2 h, 4 h, 6 h, and 24 h post-dose
Efficacy | Predose, up to 2 months post-dose
  Change in tumor size from baseline by cystoscopy, change in tumor proliferation marker Ki-67 by immunohistochemistry, change in caspase-3 expression by immunohistochemistry

CONTACTS AND LOCATIONS:
Overall Officials: Juha Peltonen, MD, Principal Investigator — CRST (Clinical Research Services Turku); Liisa Pylkkänen, MD, PhD, Study Chair — BioCis Pharma Ltd
Locations (2):
- Finland (2):
  - Tampere University Hospital, Department of Urology, Tampere
  - Turku University Hospital, Department of Surgery, Division of Urology, Turku